CLINICAL TRIAL: NCT07157644
Title: Comparison of Functional Exercise Capacity, Muscle Oxygenation, Respiratory Muscle Strength, and Physical Activity Level in Pediatric Cystic Fibrosis and Primary Ciliary Dyskinesia
Brief Title: Exercise Capacity, Muscle Oxygenation, Respiratory Muscle Strength, and Physical Activity Level in Pediatric CF and PCD
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi2707
Record Dates: First submitted 2025-08-23; First posted 2025-09-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Cystic Fibrosis (CF); Primary Ciliary Dyskinesia (PCD)
Keywords: cystic fibrosis; primary ciliary dyskinesia; muscle oxygenation; exercise tolerance; physical activity
MeSH Terms: conditions — Cystic Fibrosis; Ciliary Motility Disorders; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with Primary Ciliary Dyskinesia: Demographic information (age, gender, education level), physical characteristics (weight, height, BMI (Body Mass Index)), medical history (past and present history, family history, diagnosis, disease duration, smoking and environmental exposure, exacerbation status within the last year, number of hospital admissions and hospitalizations, medications used, parental consanguinity, socioeconomic status, number of siblings diagnosed with primary ciliary dyskinesia (PCD) or, cystic fibrosis (CF) body weight, height, and BMI Z scores were recorded. Pulmonary function, respiratory muscle strength and endurance, functional exercise capacity, muscle oxygenation, and physical activity level were assessed for all individuals.
- Patient with Cystic Fibrosis: Demographic information (age, gender, education level), physical characteristics (weight, height, BMI (Body Mass Index)), medical history (past and present history, family history, diagnosis, disease duration, smoking and environmental exposure, exacerbation status within the last year, number of hospital admissions and hospitalizations, medications used, parental consanguinity, socioeconomic status, number of siblings diagnosed with primary ciliary dyskinesia (PCD) or, cystic fibrosis (CF) body weight, height, and BMI Z scores were recorded. Pulmonary function, respiratory muscle strength and endurance, functional exercise capacity, muscle oxygenation, and physical activity level were assessed for all individuals.
- Health Controls: Demographic information (age, gender, education level), physical characteristics (weight, height, BMI (Body Mass Index)), body weight, height, and BMI Z scores were recorded. Pulmonary function, respiratory muscle strength and endurance, functional exercise capacity, muscle oxygenation, and physical activity level were assessed for all individuals.

SUMMARY:
Cystic fibrosis (CF) and primary ciliary dyskinesia (PCD) are genetic diseases characterized by chronic respiratory tract infections. In both diseases, impaired mucociliary clearance, recurrent respiratory infections, and persistent inflammation lead to progressive deterioration in respiratory function. This condition limits patients' activities of daily living, leading to physical inactivity and exercise intolerance. Functional exercise capacity in patients with CF and PCD is reduced due to increased respiratory load, musculoskeletal involvement, and nutritional deficiencies. In exercise tests involving the upper and lower extremities, both patient groups exhibited significantly lower performance compared to healthy individuals. Muscle oxygenation is particularly reduced in patients with cystic fibrosis and is associated with inadequate oxygen delivery to peripheral muscles, mitochondrial dysfunction, and increased muscle fatigue. Although studies on muscle oxygenation in PCD patients are limited, it is thought to be affected by similar pathophysiological mechanisms. Respiratory muscle strength is weakened in both patient groups due to chronic cough, hyperinflation, and increased respiratory effort. This is particularly evident in a significant decrease in inspiratory and expiratory muscle strength. The number of studies in the literature evaluating muscle oxygenation, respiratory muscle strength, and physical activity levels in patients with CF and PCD is limited. There are no studies comparing muscle oxygenation between patients with CF and PCD.

DETAILED DESCRIPTION:
In patients with cystic fibrosis (CF) and primary ciliary dyskinesia (PCD), lower extremity exercise capacity, skeletal muscle function, respiratory muscle strength, and physical activity levels are limited by various pathophysiological mechanisms. In CF patients, lower extremity exercise capacity is significantly reduced due to ventilation limitation, respiratory muscle fatigue, and mitochondrial dysfunction. Early fatigue findings such as delayed oxygen uptake and lactate accumulation have been reported in lower extremity-specific exercise tests. In PCD patients, respiratory workload increases due to ventilation-perfusion mismatch and impaired mucociliary clearance, which can limit muscle oxygen utilization during exercise. Recent studies have shown that PCD patients have lower resting muscle oxygen saturation compared to healthy individuals, but these values are relatively maintained during exercise. In CF, respiratory muscle strength is weakened, particularly at the diaphragm and intercostal muscles, leading to a decrease in ventilatory reserve during exercise. Similarly, submaximal respiratory muscle fatigue and decreased inspiratory muscle strength have been reported in patients with PCD. Regarding physical activity levels, daily activity levels in both patient groups are significantly lower than in healthy peers, and this has been associated with disease progression, muscle dysfunction, and exercise intolerance. Objectively measured studies in children and adolescents with CF have reported that they fall below the recommended daily activity level, and this inadequacy negatively impacts muscle function over time. A similar tendency toward physical inactivity is also found in PCD patients, and this is considered directly related to exercise capacity. The number of studies in the literature evaluating muscle oxygenation, respiratory muscle strength, and physical activity levels in patients with CF and PCD is limited. There are no studies comparing muscle oxygenation in patients with CF and PCD. The aim of our study was to compare functional exercise capacity, muscle oxygenation, respiratory muscle strength, and physical activity in children with CF, PCD, and healthy children.

ELIGIBILITY:
Inclusion Criteria:

Cystic fibrosis patients;

* Patients diagnosed with cystic fibrosis according to the American Cystic Fibrosis Association consensus report
* Between the ages of 6 and 18
* Clinically stable conditions

Primary ciliary dyskinesia patients;

* Patients diagnosed with primary ciliary dyskinesia according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines
* Between the ages of 6 and 18
* Clinically stable conditions

Healthy controls;

* Agreeing to participate voluntarily in the study
* Between the ages of 6 and 18

Exclusion Criteria:

Patients;

* Uncooperative
* Orthopedic or neurological disorders that will affect functional capacity
* Pneumonia or any acute infection

Healthy controls;

* Chronic disease
* Uncooperative
* Orthopedic or neurological disorders that will affect functional capacity

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Thirty-one patients with CF, 27 patients with PSD were included in the study. There are 30 healthy data.
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
Functional Exercise Capacity | First Day
  The six minute walk test (six-MWT) was used to assess functional exercise capacity. The six-MWT was administered according to the criteria of the American Thoracic Society and the European Respiratory Society. Heart rate at rest, after the test, and at the first minute of recovery were assessed using a heart rate monitor (Polar FTI00, China), blood pressure using a sphygmomanometer (Erka Perfect Aneroid, Germany), oxygen saturation using a portable pulse oximeter (Nonin Onyx Vantage 9590, Minnesota, USA), and respiratory frequency (counting the number of breaths taken per minute). The severity of dyspnea and body and leg fatigue was determined using the modified Borg Scale. The six-MWT was repeated twice. Walking distance was expressed in meters and as a percentage of the predicted value. The best walking distance result was selected for analysis. The percentage of the predicted walking distance values was calculated using the reference equation of Gibbons et al.
Muscle oxygenation (Resting muscle oxygen saturation (SmO2rest)) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the six-MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (Minimum muscle oxygen saturation (SmO2min)) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (Maximum muscle oxygen saturation (SmO2max)) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (ΔSmO2) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (SmO2averaged-min) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (SmO2averaged -max) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (ΔSmO2averaged) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (SmO2recovery) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (SmO2recovery-averaged) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (Resting total hemoglobin level (THbrest)) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded
Muscle oxygenation (Minumum total hemoglobin level (THbmin)) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6PBRT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (Maximum total hemoglobin level (Thbmax)) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (ΔTHb) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT, the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.
Muscle oxygenation (THbrecovery) | First Day
  Muscle oxygenation was assessed using the Moxy monitor device (Moxy, Fortiori Design LLC, Minnesota, ABD). During the 6MWT the device was placed on the quadriceps muscle of the dominant leg, and measurements were recorded.

SECONDARY OUTCOMES:
Heart rate | First day
  Heart rate at rest, after the test, and at the first minute of recovery were assessed using a heart rate monitor (Polar FTI00, China).
Blood pressure | First day
  Blood pressure at rest, after the test, and at the first minute of recovery were assessed using a sphygmomanometer (Erka Perfect Aneroid).
Oxygen saturation | First day
  Oxygen saturation at rest, after the test, and at the first minute of recovery were assessed using a portable pulse oximeter (Nonin Onyx Vantage 9590, Minnesota, USA).
Breathing frequency | First day
  Breathing frequency at rest, after the test, and at the first minute of recovery were assessed using a counting the number of breaths taken per minute.
Dyspnea | First day
  The severity of dyspnea was determined using the modified Borg Scale.
Body and leg fatigue | First day
  The severity of body and leg fatigue was determined using the modified Borg Scale.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function was assesed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced vital capacity (FVC) was assessed.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First Day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) was assessed.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, FEV1 / FVC was assessed.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) was assessed.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function was assessed with the spirometry. Dynamic lung volume measurements were made according to ATS and ERS criteria. With the device, peak flow rate (PEF) was assessed.
Respiratory Muscle Strength | Second Day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength were measured using a portable mouth pressure measuring device according to American Thoracic Society and European Respiratory Society criteria
Respiratory Muscle Endurance | Second Day
  Incremental threshold loading test
Physical Activity Level (Total energy expenditure) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Active energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day)) | Second day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Physical activity time (min / day)will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Average metabolic equivalent (MET / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Number of steps (steps / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Time spent lying down (min / day) days) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 4 continuous days. The patient will be informed about removing the device while taking a bath. Sleep time (min / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.

CONTACTS AND LOCATIONS:
Overall Officials: Şeyma MUTLU KAYAARSLAN, MSc, Principal Investigator — Baskent University; Meral BOŞNAK GÜÇLÜ, Prof. Dr, Study Director — Gazi University; Betül YOLERİ, MSc, Study Chair — Gazi University
Locations (1):
- Gazi University Faculty of Health Sciences Department of Cardiopulmonary Physiotherapy and Rehabilitation, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nakagomi A, Shoji T, Okada S, Ohno Y, Kobayashi Y. Validity of the augmentation index and pulse pressure amplification as determined by the SphygmoCor XCEL device: a comparison with invasive measurements. Hypertens Res. 2018 Jan;41(1):27-32. doi: 10.1038/hr.2017.81. Epub 2017 Oct 5. PMID 28978987
- [Result] Harun SN, Wainwright C, Klein K, Hennig S. A systematic review of studies examining the rate of lung function decline in patients with cystic fibrosis. Paediatr Respir Rev. 2016 Sep;20:55-66. doi: 10.1016/j.prrv.2016.03.002. Epub 2016 Mar 14. PMID 27259460
- [Result] Ratjen F, Bell SC, Rowe SM, Goss CH, Quittner AL, Bush A. Cystic fibrosis. Nat Rev Dis Primers. 2015 May 14;1:15010. doi: 10.1038/nrdp.2015.10. PMID 27189798
- [Result] Mutlu S, Bosnak Guclu M, Sismanlar Eyuboglu T, Aslan AT. Upper Extremity Exercise Capacity and Muscle Oxygenation in Patients With Primary Ciliary Dyskinesia. Pediatr Pulmonol. 2025 Jan;60(1):e27470. doi: 10.1002/ppul.27470. PMID 39785198
- [Result] Gosselink R, Troosters T, Decramer M. Peripheral muscle weakness contributes to exercise limitation in COPD. Am J Respir Crit Care Med. 1996 Mar;153(3):976-80. doi: 10.1164/ajrccm.153.3.8630582.
- [Result] Lucas JS, Barbato A, Collins SA, Goutaki M, Behan L, Caudri D, Dell S, Eber E, Escudier E, Hirst RA, Hogg C, Jorissen M, Latzin P, Legendre M, Leigh MW, Midulla F, Nielsen KG, Omran H, Papon JF, Pohunek P, Redfern B, Rigau D, Rindlisbacher B, Santamaria F, Shoemark A, Snijders D, Tonia T, Titieni A, Walker WT, Werner C, Bush A, Kuehni CE. European Respiratory Society guidelines for the diagnosis of primary ciliary dyskinesia. Eur Respir J. 2017 Jan 4;49(1):1601090. doi: 10.1183/13993003.01090-2016. Print 2017 Jan. PMID 27836958
- [Result] Sharma R, Florea VG, Bolger AP, Doehner W, Florea ND, Coats AJ, Hodson ME, Anker SD, Henein MY. Wasting as an independent predictor of mortality in patients with cystic fibrosis. Thorax. 2001 Oct;56(10):746-50. doi: 10.1136/thorax.56.10.746. PMID 11562511
- [Result] Quanjer PH, Tammeling GJ, Cotes JE, Pedersen OF, Peslin R, Yernault JC. Lung volumes and forced ventilatory flows. Report Working Party Standardization of Lung Function Tests, European Community for Steel and Coal. Official Statement of the European Respiratory Society. Eur Respir J Suppl. 1993 Mar;16:5-40. No abstract available. PMID 8499054
- [Result] de Onis M, Onyango AW, Borghi E, Siyam A, Nishida C, Siekmann J. Development of a WHO growth reference for school-aged children and adolescents. Bull World Health Organ. 2007 Sep;85(9):660-7. doi: 10.2471/blt.07.043497. PMID 18026621